CLINICAL TRIAL: NCT04749160
Title: Smart Marker Annunciating Response to Rheumatologic Treatments SMART²T
Acronym: SMART²T
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH191; 2020-A02737-32 (Other: ANSM)
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis (RA); synthetic disease modifying antirheumatic drug (csDMARD); biologic disease modifying antirheumatic drug (bDMARD); Machine Learning
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis (RA) with connected device: RA with DAS28 ≥ 3.2 despite methotrexate therapy and initiating for the first time a bDMARD or a tsDMARD.
  the physical activity and sleep quality measured with connected device
  Interventions: Device: Connected device

INTERVENTIONS:
Device: Connected device — Connected device is a smart watch (with accelerometer without location data).

SUMMARY:
European recommendations indicate to start a conventional synthetic disease modifying antirheumatic drug (csDMARD) as soon as possible to reach the remission in early RA or low disease activity in established RA. If the target is not achieved with the first csDMARD and in presence of poor prognostic, addition of a biologic (b)DMARD or a targeted synthetic (ts)DMARD should be considered . Nevertheless, as many as one-third of patients have persistent disease activity and insufficient (inadequate) response to a first b/tsDMARD according to international recommendations. This relatively long time (3 to 6 months) between treatment initiation and determination of individual clinical response represents:

* a risk for the patient who could be usually exposed to potential side effects,
* a loss of chance for the patient who will not receive an adequate treatment during the most favorable period and thus may develop irreversible lesions
* a cost for the healthcare system, especially in terms of expensive drug reimbursements, notwithstanding the increasing use of biosimilars.

Despite 20 years of research, no biomarker or no way are available in the daily practice to predict disease activity and the non-response to a b/tDMARD [11]. Thus exploration of a new approach is totally in purpose.

The aim of this project is to benefit from the declarative PRO (Patient Reported Outcomes), the physical activity and sleep quality to predict the individual clinical response to the b/tsDMARDs

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* Adult patient (over 18 years old)
* RA according to ACR/EULAR 2010 criteria since less than 6 months
* DAS28 ≥ 3.2 despite methotrexate therapy and initiating for the first time a bDMARD or a tsDMARD
* Having an internet access at home and using an email address

Exclusion Criteria:

* Other arthritis than RA
* To participate to a blind-randomized study to assess RA treatment
* Pregnancy or breastfeeding
* Patient unable to understand the study, unable to give consent
* Patient deprived of liberty or patient under guardianship
* Patient refusing to participate in the study
* Patients having difficulty using connected objects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patient with DAS28 ≥ 3.2 despite methotrexate therapy and initiating for the first time a bDMARD or a tsDMARD
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
physical activities | 3 months
  Physical activities including number of steps per day and per hour. Physical activities are measured with a smart watch (with accelerometer without location data)
physical activities and sleep quality | 3 months
  sleep quality data including time of sleeping (number of hours). sleep quality is measured with a smart watch (with accelerometer without location data)
Rapid-3 score | 3 months
  Routine Assessment of Patient Index Data (Rapid-3) score is a self-administered score demonstrated capacity to capture Rheumatoid arthritis activity (score : 0,0 to 30,0).
  Remission : score 0- 3,0 Low Disease Activity : score 3,1- 6,0 Moderate Disease Activity : score 6,1 - 12,0 High Disease Activity : score 12,1 - 30

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (13):
- France (13):
  - Centre Hospitalier de Besancon, Besançon
  - Hôpital Pellegrin, Bordeaux
  - Clinique de l'Infirmerie Protestante deLyon, Caluire-et-Cuire
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - Hôpital Sud, Grenoble
  - CH Le Mans, Le Mans
  - CHU Montpellier, Montpellier
  - Centre Hospitalier D'Orleans, Orléans
  - Hôpital Pitié Salpétrière, Paris
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Hautepierre, Strasbourg
  - Hôpital Pierre-Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No